CLINICAL TRIAL: NCT00454493
Title: The Effect of Fish Oil Supplementation on Endothelial Function, Heart Rate Variability and Intimal Media Thickness of Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Reliant Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sheba Meymandi, Director, Cardiovascular Research, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05H-561610
Record Dates: First submitted 2007-03-29; First posted 2007-03-30 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2007-03

CONDITIONS: Coronary Artery Disease
Keywords: omacor; fish oil; omega 3; fatty acids; coronary artery disease; endothelial function; heart rate variability; carotid intimal media thickness; QT dispersion
MeSH Terms: conditions — Coronary Artery Disease | interventions — Omacor

STUDY DESIGN:
Intervention Model Description: prospective, placebo-controlled, randomized, double-blind trial

ARMS (2):
- fish oil (Active Comparator)
  Interventions: Drug: Omacor (omega-3-acid ethyl esters)
- placebo (Placebo Comparator)
  Interventions: Drug: Omacor (omega-3-acid ethyl esters)

INTERVENTIONS:
Drug: Omacor (omega-3-acid ethyl esters)

SUMMARY:
The purpose of this study is to investigate whether there is a difference in endothelial function, heart rate variability and carotid intimal media thickness in patients with coronary artery disease who are receiving fish oil therapy.

One hundred patients with established coronary artery disease by coronary angiography will undergo randomization for enrollment in the study. Baseline evaluation will include assessment of brachial artery endothelial function, heart rate variability and carotid intimal media thickness. Evaluation of the endothelial function of the brachial artery will be elucidated by inflation of a blood pressure cuff around the arm for five minutes and measuring blood vessel dynamics after release of the cuff. Heart rate variability will be evaluated by 24 hour holter monitoring and analysis by standard protocol. Carotid intimal media thickness will be evaluated by ultrasound measurements guided by predetermined protocol. Patients will then be randomized to a highly purified fish oil, Omacor, 1 gram twice a day or placebo. Brachial artery ultrasound and holter monitoring will be repeated at 2 months. Carotid ultrasound will be repeated at the end of the study at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Established coronary artery disease as determined by coronary angiography within the last 5 years demonstrating at least 50% stenosis in one of the major coronary vessels
2. Age >18 and <75.

Exclusion Criteria:

1. Baseline fish oil intake ≥1g/day or fish intake >100g/day
2. Need for urgent or emergent CABG
3. Contraindication for plavix, aspirin or statin
4. Gastrointestinal malabsorption syndrome
5. Pregnancy
6. Oral contraceptive use
7. Ejection fraction <40%
8. Underlying atrial or ventricular arrhythmia
9. History of rheumatoid arthritis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percent change in flow-mediated vasodilation by brachial artery ultrasound at 2 months | 2 months
  Percent change in flow-mediated vasodilation by brachial artery ultrasound
Change in heart rate variability indices at 2 months | 2 months
  Change in heart rate variability indices on holter monitor
Percent change in carotid intimal media thickness at 12 months | 2 months
  Percent change in carotid intimal media thickness on ultrasound

SECONDARY OUTCOMES:
Change in QT dispersion interval at 2 months | 2 months
  Change in QT dispersion interval on holter monitor

CONTACTS AND LOCATIONS:
Overall Officials: Sheba K Meymandi, M.D., FACC, Principal Investigator — University of California, Los Angeles
Locations (1):
- OV-UCLA Medical Center, Sylmar, California, United States